CLINICAL TRIAL: NCT02550392
Title: Optimising Psychoeducation for Transient Ischaemic Attack and Minor Stroke Management (OPTIMISM)
Brief Title: Psychoeducation for Transient Ischaemic Attack and Minor Stroke
Acronym: OPTIMISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: The Stroke Association, United Kingdom (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15079; TSA PDF 2015-01 (Other Grant/Funding Number: Stroke Association)
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Transient Ischaemic Attack; Stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group psychoeducation (Experimental): The intervention group will receive a group psychoeducational intervention (designed in Phase 1: Qualitative study) and usual care.
  Interventions: Behavioral: Psychoeducation
- Control group (No Intervention): Participants in the usual care control group will continue to receive all other services routinely available to them as is usual practice.

INTERVENTIONS:
Behavioral: Psychoeducation — A time-limited group psychoeducational intervention that will aim to offer educational, psychological and social support.
  Arms: Group psychoeducation

SUMMARY:
Transient Ischaemic Attack (TIA), also called 'ministroke' is characterised by shortlasting symptoms that generally do not cause permanent damage. 'Minor stroke' is a term used to describe a stroke with mild and nondisabling symptoms. TIA and minor stroke patients account for more than half of all cases of stroke and they are at a higher risk to suffer a major stroke. Currently, management of TIA/minor stroke patients is mainly focused on identifying and reducing risk factors for a later stroke. However, people after a TIA often have limited access for further specialist support from stroke-specific rehabilitation services. Although there is variability in the level of recovery and severity of symptoms after TIA and minor stroke, there is evidence that these patients may experience difficulties that affect their quality of life including anxiety and depression.

This study aims to develop, tailor and target the delivery of a time-limited group intervention that offers educational, psychological and social support for people following TIA and minor stroke. A qualitative study (Phase 1) will be conducted with service users and experts working with people with TIA/minor stroke to develop the psychoeducational intervention. Following this, we will conduct a feasibility randomised controlled trial in one centre (Phase 2) to explore whether this group psychoeducational intervention for people after TIA and minor stroke carers is acceptable and to determine the feasibility of the proposed evaluation and the sample size needed in a definite trial.

DETAILED DESCRIPTION:
Participants will complete measures at baseline and then randomly allocated to receive the intervention or usual care. The intervention group will receive a group psychoeducational intervention (designed in Phase 1: Qualitative study) in addition to self-help leaflets and usual care. It is anticipated that the intervention will be offered in 6 two-hour sessions over 3 months by an assistant psychologist. The control group will receive usual care plus self-help leaflets on relevant topics. All participants will complete outcome measures at 3 and 6 months after randomisation. We will test the feasibility, tolerability and acceptability of delivering the intervention and will record data on study completion and attrition. Findings will inform the development of a larger trial and will determine if the content and delivery of the intervention meets the needs of people after TIA and minor stroke.

ELIGIBILITY:
Inclusion criteria:

* adults with a first/recurrent TIA or minor stroke;
* identified within 6 months of their diagnosis;
* who are independent with activities of daily living;
* who consent to take part

Exclusion criteria:

* diagnosis of dementia;
* receiving psychological interventions for mental health difficulties immediately prior to their TIA/minor stroke, visual or hearing impairments that would impact on ability to complete baseline assessments;
* cognitive or communication difficulties that would impact on ability to complete baseline assessments and to participate in group sessions;
* unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited to the trial | up to 1 year
Number of participants who completed the trial | participants will be followed for the duration of the trial, an expected average of 12 months

SECONDARY OUTCOMES:
Mood | baseline, 3 and 6 months follow-up
  General Health Questionnaire-30 (GHQ-30)
Health-related Quality of Life | baseline, 3 and 6 months follow-up
  EuroQuol-5D
Knowledge and Satisfaction | baseline, 3 and 6 months follow-up
  Knowledge and Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eirini Kontou, PhD DClinPsy, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No